CLINICAL TRIAL: NCT01272622
Title: KRANIOPHARYNGEOM 2007 - Multicenter Prospective Study of Children and Adolescents With Craniopharyngioma
Brief Title: Prospective Study of Children and Adolescents With Craniopharyngioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinikum Oldenburg gGmbH (Other)
Collaborators: German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other); Arbeitsgemeinschaft Pädiatrische Endokrinologie (APE) (Unknown); Deutsche Gesellschaft für Endokrinologie (DGE) (Unknown); Arbeitsgemeinschaft Pädiatrische Radioonkologie (APRO) (Unknown); Deutsche Gesellschafr für Radioonkologie (DEGRO) (Unknown); Deutsche Kinderkrebsstiftung (Other); International Society of Paediatric Oncology (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Hermann Mueller, Professor MD, Klinikum Oldenburg gGmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DKSR 463
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Craniopharyngioma; Obesity
Keywords: Quality of life; Endocrinology; Oncology; Hypothalamus; Irradiation; Neurosurgery; Pediatric Brain tumors; Randomized trial
MeSH Terms: conditions — Craniopharyngioma; Obesity; Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Other): Children and adolescents >= 18 years of age new diagnosed with craniopharyngioma
  * >= 5 years of age and with incomplete resected tumor => randomized in two arms: immediate irradiation after surgery
  Interventions: Radiation: Radiation
- Arm II (Other): incomplete resection, wait and watch, MRI-controls every 3 months, and irradiation at the time of progression of residual tumor
  Interventions: Other: wait and watch

INTERVENTIONS:
Radiation: Radiation — Immediate irradiation after incomplete resection (fractionated, percutaneous irradiation, 54 gy)
  Arms: Arm I
Other: wait and watch — wait ans watch, MRI controls, irradiation at the time of progression of residual tumor
  Arms: Arm II

SUMMARY:
The present investigation is a prospective, multicenter study evaluating craniopharyngioma patients' prognoses following the various currently-practiced therapeutic strategies.Primary goals of the study are to establish quality standards and compare the various therapy strategies with respect to their effectiveness and impact on the quality of life of treated patients. A stratified randomization of two treatment arms will be conducted with respect to timing of postoperative irradiation for the subgroup of patients ≥5 years of age whose tumors are incompletely resected. The researchers will investigate whether an immediate, postoperative irradiation is superior to progression-contingent irradiation based on alterations to quality of life (PEDQOL) from the time randomization is initiated (3rd month post op) to 3 years after randomization. Progression-free survival and overall survival will be examined as closely-related subgoals.Postoperative data will be evaluated via a surveillance study for all complete resection patients as well as for those patients under 5 years of age regardless of their resection grade.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with craniopharyngioma for the first time
2. Age at diagnosis 18 years or less of age
3. Agreement from patient's parents or legal guardian as well as the patient

Criteria for inclusion in randomization study

1. Histological diagnosis of craniopharyngioma
2. Age at diagnosis 18 years or less of age
3. Age at primary surgery over 5 years of age
4. Incomplete primary resection
5. Reference radiological confirmation of an incomplete resection
6. Agreement from patient's parents or legal guardian as well as the patient

Exclusion Criteria:

Age at diagnosis over 18 years of age No QoL measurement for randomization (3 months after surgery).

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2007-10; Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Quality of life | 3 years after diagnosis
  •Randomized investigation of children (≥ 5 years of age) and adolescent QoL changes (main goal assessment) following incomplete craniopharyngioma resections at primary diagnosis per QoL endpoint scores (PEDQOL "physical functions" domain) measured from 3rd month after surgery for 3 years after randomization; and the progression-free and total survival rates (subgoal assessments) relative to how these rates relate to postoperative irradiation timing (immediate postsurgery irradiation versus wait-and-see approach + progression-contingent irradiation of residual tumor).

SECONDARY OUTCOMES:
Rate of Progression or relapse | 3 years after surgery
  * Compilation of applied therapy strategies for craniopharyngiomas in children and adolescents using data capture conforming to SIOP brain tumor groups
  * Evaluation of patients' remission status following the various therapy strategies/modalities for craniopharyngiomas using data detection consistent with SIOP brain tumor groups
  * Evaluation of the health status (ophthalmologic, neuropsychologic and endocrine conditions) and health-related QoL of children and adolescents following treatment of craniopharyngiomas using data capture conforming to SIOP brain tumor groups

CONTACTS AND LOCATIONS:
Overall Officials: Hermann L Müller, MD, Principal Investigator — Klinikum Oldenburg gGmbH
Locations (1):
- Klinikum Oldenburg, Oldenburg, Lower Saxony, Germany

REFERENCES:
- [Derived] Sowithayasakul P, Beckhaus J, Ozyurt J, Bison B, Friedrich C, Muller HL. Prolactin serum concentrations in childhood-onset craniopharyngioma patients. J Endocrinol Invest. 2025 Sep;48(9):2041-2051. doi: 10.1007/s40618-025-02622-4. Epub 2025 Jun 7. PMID 40481916
- [Derived] Mann-Markutzyk LV, Beckhaus J, Ozyurt J, Mehren A, Friedrich C, Muller HL. Daytime sleepiness and health-related quality of life in patients with childhood-onset craniopharyngioma. Sci Rep. 2025 Mar 19;15(1):9407. doi: 10.1038/s41598-025-94384-5. PMID 40108339
- [Derived] Friedrich C, Boekhoff S, Bischoff M, Beckhaus J, Sowithayasakul P, Calaminus G, Eveslage M, Valentini C, Bison B, Harrabi SB, Krause M, Timmermann B, Muller HL. Outcome after proton beam therapy versus photon-based radiation therapy in childhood-onset craniopharyngioma patients-results of KRANIOPHARYNGEOM 2007. Front Oncol. 2023 Oct 27;13:1180993. doi: 10.3389/fonc.2023.1180993. eCollection 2023. PMID 37965466
- [Derived] Sowithayasakul P, Beckhaus J, Boekhoff S, Friedrich C, Calaminus G, Muller HL. Vision-related quality of life in patients with childhood-onset craniopharyngioma. Sci Rep. 2023 Nov 10;13(1):19599. doi: 10.1038/s41598-023-46532-y. PMID 37949931
- [Derived] Wagener K, Beckhaus J, Boekhoff S, Friedrich C, Muller HL. Sporadic and neurofibromatosis type 2-associated meningioma in children and adolescents. J Neurooncol. 2023 Jul;163(3):555-563. doi: 10.1007/s11060-023-04344-0. Epub 2023 Jul 4. PMID 37402092
- [Derived] Beckhaus J, Friedrich C, Boekhoff S, Calaminus G, Bison B, Eveslage M, Timmermann B, Flitsch J, Muller HL. Outcome after pediatric craniopharyngioma: the role of age at diagnosis and hypothalamic damage. Eur J Endocrinol. 2023 Mar 2;188(3):lvad027. doi: 10.1093/ejendo/lvad027. PMID 36857103
- [Derived] Boekhoff S, Bison B, Eveslage M, Sowithayasakul P, Muller HL. Craniopharyngiomas presenting as incidentalomas: results of KRANIOPHARYNGEOM 2007. Pituitary. 2019 Oct;22(5):532-541. doi: 10.1007/s11102-019-00983-7. PMID 31440945
- [Derived] Daubenbuchel AM, Hoffmann A, Eveslage M, Ozyurt J, Lohle K, Reichel J, Thiel CM, Martens H, Geenen V, Muller HL. Oxytocin in survivors of childhood-onset craniopharyngioma. Endocrine. 2016 Nov;54(2):524-531. doi: 10.1007/s12020-016-1084-5. Epub 2016 Sep 1. PMID 27585663
- [Derived] Hoffmann A, Warmuth-Metz M, Lohle K, Reichel J, Daubenbuchel AM, Sterkenburg AS, Muller HL. Fusiform dilatation of the internal carotid artery in childhood-onset craniopharyngioma: multicenter study on incidence and long-term outcome. Pituitary. 2016 Aug;19(4):422-8. doi: 10.1007/s11102-016-0722-5. PMID 27125511